CLINICAL TRIAL: NCT06008912
Title: Investigation of the Effect of Calisthenic Exercise Training Combined With Aerobic Exercise on Exercise Tolerance, Physical Fitness and Plasma Lipid Profile in Patients With Dyslipidemia
Brief Title: Effect of Calisthenic Exercise Training Combined With Aerobic Exercise in Patients With Dyslipidemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Furkan Özdemir, Lecturer, Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KA-22027
Record Dates: First submitted 2023-08-08; First posted 2023-08-24 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Dyslipidemias
Keywords: Dyslipidemia; Calisthenic Exercise; Exercise Capacity
MeSH Terms: conditions — Dyslipidemias | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Experimental model of study consist from three arm.
  * First Arm: Patients will take aerobic exercise training in 3 days per week, and 7 days per week calisthenic exercises for upper extremity, lower extremity and trunk, for 8 weeks.
  * Second Arm: Patients will take aerobic exercise training in 3 days per week, for 8 weeks.
  * Third Arm: Patients will take physical activity recommendations, and just screening after 8 weeks.
Who Masked: Participant, Care Provider
Masking Description: Patients and his/her caregivers will allocate in study via computer based randomisation, and will not know about his/her and also other participants group in study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Calisthenic + Aerobic Exercise Group (Experimental): Patients will take aerobic exercise training in 3 days per week, and 7 days per week calisthenic exercises for upper extremity, lower extremity and trunk, for 8 weeks.
  Interventions: Other: Calisthenic Exercises; Other: Aerobic Exercises
- Aerobic Exercise Group (Active Comparator): Patients will take aerobic exercise training in 3 days per week, for 8 weeks.
  Interventions: Other: Aerobic Exercises
- Control Group (No Intervention): Patients will take physical activity recommendations, and just screening after 8 weeks.

INTERVENTIONS:
Other: Calisthenic Exercises — Exercises for upper extremity, lower extremity and trunk which applying just patient's own body weight via using body mechanics. There is no need for any tools for exercises.
  Arms: Calisthenic + Aerobic Exercise Group
Other: Aerobic Exercises — Exercises which loading cardiovascular, respiratory and muscular system at the same time. Treadmill training will apply in the study.
  Arms: Aerobic Exercise Group; Calisthenic + Aerobic Exercise Group

SUMMARY:
Dyslipidemia is expressed as the serum concentration of lipid molecules with different structures outside the normal level. Deviation of serum lipid level from normal is accepted as the primary or most important factor in various cardiac and metabolic diseases, especially atherosclerosis. Dyslipidemia-related cardiovascular structure change is accepted as an important public health problem worldwide, and it is stated that the combined use of medical treatment, changes in diet and physical activity/structured exercise programs in the treatment of dyslipidemia is important in the success of treatment.

DETAILED DESCRIPTION:
Lipid profile disorders (especially high total blood cholesterol level) are a major problem worldwide, and accepted as a important public health problem. It has been reported that approximately one out of every three people worldwide has been exposed to dyslipidemia risk factors. Prevalence studies showed that lipid profile disorders vary between 6.9% and 43.6% worldwide. Today, ischemic heart and central nervous system diseases are the most important causes of mortality and morbidity in adult population, globally. Especially, it is accepted that lipid profile disorders are the leading risk factors causing ischemic heart diseases.

Prevalence varies according to regions, lifestyle habits and individual factors, because of lipid profile disorders are caused by many different genetic and environmental factors. Apart from individual factors, there are other factors that lipid weight in diet, nutrient deficiencies which balancing lipid metabolism, physical activity level and inactivity, other comorbid diseases, and medical treatments change lipid metabolism in individuals and lead to deterioration in lipid profile. Especially lifestyle habits affect lipid metabolism most easily and they are the most easily modifiable factors.

It is recommended to apply a multi-dimensional approach when treating lipid profile disorders. It is recommended that, to include diet counseling and exercise therapy in these approaches. Exercise therapy is especially recognized as an important treatment option for the control and treatment of obesity, hypertension, hyperglycemia and metabolic syndrome symptoms that may accompany dyslipidemia.

It has been reported that aerobic exercise programs increase patients' quality of life and functionality which applied to dyslipidemia patients, but there is lack of information available in literature about the effects of calisthenic exercises in patients with dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Screening by the internal medicine clinic with the diagnosis of dyslipidemia
* Being between 18 to 65 years old
* Volunteering to participate in the research

Exclusion Criteria:

* Having any cardiac disease
* Having a co-existing psychiatric illness (like schizophrenia, bipolar disorder, etc.)
* Being infected with COVID-19 in the last 3 months
* Having any neurological problems that may affect cooperation
* Having pulmonary or orthopedic problem that may affect functional capacity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-05-14 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Exercise Capacity | Second Day
  Cardiopulmonary exercise capacity will assess as primary outcome measure, via cardiopulmonary exercise test (CPET).

SECONDARY OUTCOMES:
Blood Lipids Concentration Assessment | First Day
  Concentration of LDL-C, HDL-C, Total cholesterol (TC) and Triglyceride (TG) will assess in blood (in mg/dL units of measure) after 12 hours fasting.
Apolipoprotein A1 Concentration Assessment | First Day
  Concentration of Apolipoprotein A1 will assess in blood (in g/dL units of measure) after 12 hours fasting.
Blood Sugar Concentration Assessment | First Day
  Concentration of fasting blood sugar (in mmol/L units of measure) and rate of HbA1c (in % units of measure) will assess in blood after 12 hours fasting.
C-reactive Protein Concentration Assessment | First Day
  Concentration of C-reactive protein (in mg/dL units of measure) will assess in blood after 12 hours fasting.
Sit-to-Stand Test | First Day
  A one-minute sit-to-stand test will be applied to the patients. One standing position followed by sitting will count as one cycle. Patients' total cycles within 60 seconds will be counted as test score (in cycle/minute units of measure)
Timed Up-and-Go Test | First Day
  Timed up-and-go test will be applied to the patients. Patients will be asked to get up from the chair, walk the 3-meter distance, return and sit back in the chair, as quickly as possible. The total time that patients complete the test and sit on the chair again will be recorded as the test score (in second/lap units of measure).
Peripheral Muscle Strength Assessment | First Day
  The muscle strength of the shoulder abductor and knee extensor muscles on the dominant and non-dominant sides of the patients will be evaluated with a portable dynamometer. During the evaluations, the patients will be asked to try to resist the force to be applied in the opposite direction of the relevant muscle's function with isometric muscle contraction. The force released during the test will be measured and the highest score (in newton [N] units of measure) will be recorded for each muscle within 3 tests.
Hand-Grip Strength Assessment | First Day
  The hand grip strength of the patients will be measured with a portable hand dynamometer. The patients will be asked to grasp the dynamometer with their fingers on the dominant and non-dominant side and squeeze it most strongly. The highest score (in kilogram force [KgF] units of measure) of 3 measurements on both sides will be recorded.
Flexibility Assessment | First Day
  Flexibility of patients will be evaluated with sit-and-reach test. Patients will be asked to stretch their hands on a bench with a measuring ruler while in a long sitting position with the ankle angled at 90 degrees and the knee fully extended. How many centimeters ahead or behind the toes of the patient's fingertips will be measured.

OTHER OUTCOMES:
Quality of Life Assessment | Second Day
  Quality of life will assess via Short Form-36 Quality of Life Questionnaire. The questionnaire consist from 36 questions and total score ranges between 0 to 100 point. Higher scores shows better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2015 Risk Factors Collaborators. Global, regional, and national comparative risk assessment of 79 behavioural, environmental and occupational, and metabolic risks or clusters of risks, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1659-1724. doi: 10.1016/S0140-6736(16)31679-8. PMID 27733284
- [Background] Rivas-Gomez B, Almeda-Valdes P, Tussie-Luna MT, Aguilar-Salinas CA. DYSLIPIDEMIA IN MEXICO, A CALL FOR ACTION. Rev Invest Clin. 2018;70(5):211-216. doi: 10.24875/RIC.18002573. PMID 30307444
- [Background] Pan L, Yang Z, Wu Y, Yin RX, Liao Y, Wang J, Gao B, Zhang L; China National Survey of Chronic Kidney Disease Working Group. The prevalence, awareness, treatment and control of dyslipidemia among adults in China. Atherosclerosis. 2016 May;248:2-9. doi: 10.1016/j.atherosclerosis.2016.02.006. Epub 2016 Feb 27. PMID 26978581
- [Background] Zhang M, Deng Q, Wang L, Huang Z, Zhou M, Li Y, Zhao Z, Zhang Y, Wang L. Prevalence of dyslipidemia and achievement of low-density lipoprotein cholesterol targets in Chinese adults: A nationally representative survey of 163,641 adults. Int J Cardiol. 2018 Jun 1;260:196-203. doi: 10.1016/j.ijcard.2017.12.069. PMID 29622441
- [Background] Yang F, Ma Q, Ma B, Jing W, Liu J, Guo M, Li J, Wang Z, Liu M. Dyslipidemia prevalence and trends among adult mental disorder inpatients in Beijing, 2005-2018: A longitudinal observational study. Asian J Psychiatr. 2021 Mar;57:102583. doi: 10.1016/j.ajp.2021.102583. Epub 2021 Feb 5. PMID 33581368
- [Background] GBD 2019 Diseases and Injuries Collaborators. Global burden of 369 diseases and injuries in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2020 Oct 17;396(10258):1204-1222. doi: 10.1016/S0140-6736(20)30925-9. PMID 33069326
- [Background] Tietge UJ. Hyperlipidemia and cardiovascular disease: inflammation, dyslipidemia, and atherosclerosis. Curr Opin Lipidol. 2014 Feb;25(1):94-5. doi: 10.1097/MOL.0000000000000051. No abstract available. PMID 24398450
- [Background] Villarreal-Molina MT, Aguilar-Salinas CA, Rodriguez-Cruz M, Riano D, Villalobos-Comparan M, Coral-Vazquez R, Menjivar M, Yescas-Gomez P, Konigsoerg-Fainstein M, Romero-Hidalgo S, Tusie-Luna MT, Canizales-Quinteros S; Metabolic Study Group. The ATP-binding cassette transporter A1 R230C variant affects HDL cholesterol levels and BMI in the Mexican population: association with obesity and obesity-related comorbidities. Diabetes. 2007 Jul;56(7):1881-7. doi: 10.2337/db06-0905. Epub 2007 Feb 7. PMID 17287470
- [Background] Villarreal-Molina MT, Flores-Dorantes MT, Arellano-Campos O, Villalobos-Comparan M, Rodriguez-Cruz M, Miliar-Garcia A, Huertas-Vazquez A, Menjivar M, Romero-Hidalgo S, Wacher NH, Tusie-Luna MT, Cruz M, Aguilar-Salinas CA, Canizales-Quinteros S; Metabolic Study Group. Association of the ATP-binding cassette transporter A1 R230C variant with early-onset type 2 diabetes in a Mexican population. Diabetes. 2008 Feb;57(2):509-13. doi: 10.2337/db07-0484. Epub 2007 Nov 14. PMID 18003760
- [Background] De Sousa SM Dr, Norman RJ Prof. Metabolic syndrome, diet and exercise. Best Pract Res Clin Obstet Gynaecol. 2016 Nov;37:140-151. doi: 10.1016/j.bpobgyn.2016.01.006. Epub 2016 Feb 10. PMID 26972165
- [Background] Wang Y, Xu D. Effects of aerobic exercise on lipids and lipoproteins. Lipids Health Dis. 2017 Jul 5;16(1):132. doi: 10.1186/s12944-017-0515-5. PMID 28679436
- [Background] Miles L. Physical activity and health. Nutr Bull [Internet]. 2007 Dec;32(4):314-63. Available from: http://doi.wiley.com/10.1111/j.1467-3010.2007.00668.x
- [Background] Strunk RC, Mrazek DA, Fukuhara JT, Masterson J, Ludwick SK, LaBrecque JF. Cardiovascular fitness in children with asthma correlates with psychologic functioning of the child. Pediatrics. 1989 Sep;84(3):460-4. PMID 2771549
- [Background] Carson KV, Chandratilleke MG, Picot J, Brinn MP, Esterman AJ, Smith BJ. Physical training for asthma. Cochrane Database Syst Rev. 2013 Sep 30;2013(9):CD001116. doi: 10.1002/14651858.CD001116.pub4. PMID 24085631
- [Background] Eime RM, Young JA, Harvey JT, Charity MJ, Payne WR. A systematic review of the psychological and social benefits of participation in sport for children and adolescents: informing development of a conceptual model of health through sport. Int J Behav Nutr Phys Act. 2013 Aug 15;10:98. doi: 10.1186/1479-5868-10-98. PMID 23945179
- [Derived] Ozdemir F, Saglam M, Aksel Uylar AA, Uyaroglu OA, Basaran NC, Tanriover MD, Yagli NV. Could calisthenic exercises improve maximal exercise capacity, peripheral muscle strength and quality of life in dyslipidemia? PLoS One. 2025 Jun 17;20(6):e0326026. doi: 10.1371/journal.pone.0326026. eCollection 2025. PMID 40526594